CLINICAL TRIAL: NCT02127359
Title: CanSeq: Whole-Exome Sequencing (WES) of Cancer Patients
Brief Title: Whole-Exome Sequencing (WES) of Cancer Patients
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nikhil Wagle, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 12-078
Record Dates: First submitted 2013-02-19; First posted 2014-04-30 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Lung Adenocarcinoma; Colon Adenocarcinoma
Keywords: Metastatic
MeSH Terms: conditions — Adenocarcinoma of Lung; Colonic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung/Colon Adenocarcinomas: Metastatic lung and colon adenocarcinomas

SUMMARY:
Cancers occur when the molecules that control normal cell growth (genes and proteins) are altered. Changes in the tumor genes and in the genes of normal cells are called "alterations." Many of these alterations can be detected by directly examining cancer cells in a tumor or circulating in blood. Several alterations that occur repeatedly in certain types of cancers have already been identified. These discoveries ahve led to the development of new drugs that "target" those alterations. More remain to be discovered.

Some of the alterations are found in genes. Genes are composed of DNA "letters," which contain the instructions that tell the cells in our bodies how to grow and work. Genes make proteins which actually carry out the instructions in our cells.

We would like to use your DNA to look for alterations in the genes in cancer cells and blood cells using a technology called "sequencing." Gene sequencing is a way of reading the DNA to identify errors in genes that may contribute to the behavior of cells. Some changes in genes occur only in cancer cells. Others occur in normal cels as well, in the genes that may have been passed from parent to child. This research study will examine both kinds of genes.

The purpose of this research study is to perform gene sequencing (gene tests) on your cancer cells (obtained from biopsies or surgery) and normal tissues (usually blood). The results of the gene tests will be used to try to develop better ways to treat and prevent cancers. We will also study better ways to communicate the results of these complex gene tests to you and your doctors, and to help you and your doctors use this information to choose the best paths for treatment. As part of this work, we may also learn things about the genes in your normal cells; some of that information will also be shared wtih you and your doctors if you so choose.

Importantly, this study will use tissue specimens that have already been collected and stored in the pathology department as part of your clinical care or as part of other research studies you may be participating in. In this study, gene tests will be performed on material only after the necessary clinical tests have been performed. In general, no additional invasive procedures will be required.

DETAILED DESCRIPTION:
If you agree to take part in this study, we are asking your permission to obtain an additional sample of blood (2 tubes or 4 teaspoons). Cells from the blood contain normal, non-cancer cell DNA which is needed for the analysis.

One of the main reasons to study the genetic characteristics of cancers is to learn whether they can predict response to existing treatments. Therefore, in this study, we would also link the results of gene tests on your cancer wtih medical information that has been generated during the course of your treatment. The medical information is contained in your medical record.

A small number of the gene test results may have importance for your health or treatment. For example, they might uncover gene alterations known to make cancers respond to (or be resistant to) specific therapies. Therefore, we are asking you to consider whether or not you would like us to inform your doctor and you about some of the results of these gene tests.

Your doctor may contact you about results of gene tests, but only if the results could impact your cancer treatment or other disease directly, or if you have given your permission for him or her to do so. In some cases, a research doctor may contact you to find out if you would be interested in participating in a different research study based on information thay may have been found in your tissue or blood samples, or in your survey/interview responses. We will also ask you to provide the name and contact information for a relative who may know your whereabouts, or who could decide about using your information for research in the future, if you are not available to give permission yourself.

Some of your specimens, as well as some of the material generated during the analysis of your tissues or blood, may be useful for study in the future, with newer technologies and approaches. We are asking your permission to store these specimens and materials in a secure biologic sample storage facility for possible later research.

We are also asking you to participate in two surveys related to the study at a few time points. These time points include when you first join the study, and after you receive any results from the gene tests done on your samples. The surveys seek to learn how you are thinking about this type of genetic analysis, and the ways in which the information can be shared with you that would be most helpful.

Some study participants will also be invited to take part in study-related interviews. The purpose of these interviews is to understand what you expect will happen as a result of the gene tests, and how the results of the gene tests may have affected you.

The surveys should take no more than 15 minutes to complete. The interviews are expected to take approximately 45 minutes to complete.

Finally, rapid progress in understanding and treating cancer will occur when some of the genetic information derived from your tissues and blood can be shared with other researchers. In particular, the National Institutes of Health (NIH) and other organizations have developed special data (information) repositories that analyze data and collect the results of certain types of genetic studies. These central banks will store your genetic information, samples, and survey/interview information and provide them to qualified researchers to do more studies. Therefore, we are also asking your permission to share your results with these special banks. Your information or samples will be sent only with a code number attached. Your name or other directly identifiable information will not be shared with data banks or other investigators. There are many safeguards in place to protect your information and samples while they are stored in repositories and used for research. although there may be a slight risk of loss of privacy when sharing this information with these banks, we have established procedures to encode your samples and information and protect your data. Although we will do everything we can to protect the privacy of your data, we cannot absolutely guarantee its privacy or predict how genetic information will be used in the future.

ELIGIBILITY:
Inclusion Criteria:

* Have previously consented to DF/HCC Protocol 11-104, 02-180 and/or are currently receiving clinical testing for KRAS mutations at BWH
* Have a diagnosis of advanced lung or colorectal adenocarcinoma
* Life expectancy of at least 6 months
* Sufficient genomic DNA available for whole exome sequencing and CLIA validation
* Have a treating oncologist who is participating in the physician study
* Speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dana-Farber Cancer Institute patients who are identified as oncology patients or patients suspected to have an eligible cancer diagnosis as defined by their providers.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2012-09; Primary Completion 2017-04 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of WES in Cancer patients | 2 years
  To implement a production-scale platform for whole exome sequencing from archival (FFPE) material. To obtain tumor and germline specimens from patients with metastatic cancer who are receiving treatment at Dana-Farber Cancer Institute, beginning with metastatic lung and colon adenocarcinomas. To perform whole exome sequencing on these specimens in order to determine somatic and germline genomic alterations that may be relevant to the development or treatment of cancer. To develop and implement an analytical and interpretive framework to prioritize clinically important genomic alterations.
Clinical Impact of Whole Exome Sequencing in Cancer Patients | 2 years
  To determine the clinical impact of somatic and germline whole exome sequencing in cancer patients. To determine the feasibility of whole exome sequencing of clinical cancer patients with advanced solid tumors, beginning with lung and colon adenocarcinomas. To establish a system of review and disclosure of results, including selected incidental results unrelated to the patients' cancer diagnoses, to physicians, patients and their families. To describe the impact of whole exome sequencing data on the medical management of patients with advanced solid tumors.
Describe Impact of Information Derived from Exome Sequencing | 2 years
  To describe the impact of information derived from somatic and germline whole-exome sequencing (WES) on cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Wagle, MD, Principal Investigator — Dana-Farber Cancer Insitute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Insitute, Boston, Massachusetts

REFERENCES:
- [Derived] Gray SW, Park ER, Najita J, Martins Y, Traeger L, Bair E, Gagne J, Garber J, Janne PA, Lindeman N, Lowenstein C, Oliver N, Sholl L, Van Allen EM, Wagle N, Wood S, Garraway L, Joffe S. Oncologists' and cancer patients' views on whole-exome sequencing and incidental findings: results from the CanSeq study. Genet Med. 2016 Oct;18(10):1011-9. doi: 10.1038/gim.2015.207. Epub 2016 Feb 11. PMID 26866579